CLINICAL TRIAL: NCT06148376
Title: Application of a Protocol of Personalized Medicine in Patients With Type 2 Diabetes Mellitus and Multiple Doses of Insulin in Routine Clinical Care
Acronym: POMA
Status: Recruiting | Type: Observational
Sponsor: Hospital Arnau de Vilanova (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Marta Hernandez Garcia, MD PhD, Hospital Arnau de Vilanova
Other Study IDs: 2965LO
Record Dates: First submitted 2023-11-18; First posted 2023-11-28 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes Mellitus; Multiple Dose Insulin Therapy
Keywords: Type 2 Diabetes Meliitus; Multiple dose insulin therapy; personalized medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDI T2DM: Patients wit type 2 diabetes (T2DM) treated with multiple dose insulin therapy (MDI)
  Interventions: Other: Personalized treatment

INTERVENTIONS:
Other: Personalized treatment — Discontinue prandial insulin treatment

SUMMARY:
The goal of this observational study is to test a protocol of personalized medicine in routine clinical practice in people with type 2 diabetes (T2DM) treated with multiple dose insulin injections (MDI).

The main question[s] it aims to answer are:

• Are c-peptide titers and B-cell autoimmunity useful to help the decision of suspending prandial insulin in patients with T2DM treated with MDI?

Participants will:

* Wear a continuous glucose monitor for 10-14 days
* Will be asked for a C-peptide and GAD antibody test (GADA)
* Will stop prandial insulin and switch to other diabetes treatments if needed if c-peptide is > 0.7 mmol/L and/or C-peptide is > 0.3 mmol/L and GADA are negative
* Will be followed-up by their GP in routine clinical practice
* Will be assessed after 6 months (CGM, HbA1c, quality of life (QoL)

DETAILED DESCRIPTION:
An algorithm will be applied in which, depending on the presence/absence of pancreatic autoimmunity and the estimation of pancreatic reserve, the same treatment will be maintained and CGM (continuous glucose monitoring) will be initiated or the prandial insulin and the treatment will be adjusted following the main clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with multiple dose insulin therapy

Exclusion Criteria:

* Gestation or planning gestation in the following 12 months
* Glucocorticoid use for an acute condition
* Transient insulinisationt (less than 6 months)
* Any condition that prevents the patient or their caregiver from following up for 6 months
* Severe mental illness
* Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients in our territory treated with multiple dose insulin therapy without exclusion criteria are elegible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients whose prandial insulin is withdrawn | At 6 months from the inclusion
  Percentage of patients whose prandial insulin is withdrawn

SECONDARY OUTCOMES:
Glucose control | 6 months
  HbA1c, continuous glucose monitoring data
Number of severe hypoglycaemia events | 6 months
  Severe hypoglycemia defined in Seaquist ER, Anderson J, Childs B, et al. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013;36(5):1384-1395.
Diabetes quality of life | 6 months
  ESDQoL
Adherence to trearment | 6 months
  ARMS-E questionnaire
Diabetes treatment satisfaction | 6 months
  DTSQs, DTSQc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marta Hernández, MD PhD, Principal Investigator — Hospital Arnau de Vilanova
Locations (2):
- Spain (2):
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Centres Atenció Primària Lleida, Alt Pirineu i Aran, Lleida

IPD SHARING:
Plan to Share IPD: No